CLINICAL TRIAL: NCT02540967
Title: Drug Use Investigation of Gadovist
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17512
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Magnetic Resonance Imaging; Image Enhancement
Keywords: Contrast enhancement in the following MR imaging; Brain and spine; Body and extremities; Gadobutrol
MeSH Terms: interventions — gadobutrol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BAY86-4875: Gadovist administration goup
  Interventions: Drug: Gadobutrol (Gadavist/Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadavist/Gadovist, BAY86-4875) — Gadovist dosage following summary of product characteristics

SUMMARY:
The objectives of this study are to investigate the safety and effectiveness of Gadovist.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, continuous submission safety study that includes patients who planned Gadolinium (Gd) contrast enhanced Magnetic Resonance Imaging (MRI) in accordance with approved label. The investigator will have made the choice of Gd enhanced MRI (the decision to use Gadovist according the Japanese Package Insert prior to enrolling the patient in this study).

The study period is 3 years. Data analysis period is 1 year. In total, 3300 patients will be recruited.

For each patient, data are collected as defined in the case report form (CRF) at the visit for MRI examination (as per investigators routine practice).

ELIGIBILITY:
Inclusion Criteria:

* Patients who perform contrast enhanced Magnetic Resonance Imaging (MRI) with Gadovist.

Exclusion Criteria:

* Patients who are contraindicated based on approved label.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female and male patients who planned Gd contrast enhanced MRI in accordance with approved label. Eligible patients who receive Gadovist will be enrolled and documented in the eCRF
Sampling Method: Non-Probability Sample
Enrollment: 3357 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Number of episodes of adverse events as a measure of safety and tolerability | Up to 3 days

SECONDARY OUTCOMES:
Number of episodes of adverse drug reactions and adverse events | Up to 3 days
  In subpopulations
Contrast enhancement | At the time of MRI
  Investigator Discretion as very improved , improved, not changed, degraded, not evaluable.
  MRI- Magnetic Resonance Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, Japan

REFERENCES:
- [Result] Tsushima Y, Awai K, Shinoda G, Miyoshi H, Chosa M, Sunaya T, Endrikat J. Post-marketing surveillance of gadobutrol for contrast-enhanced magnetic resonance imaging in Japan. Jpn J Radiol. 2018 Nov;36(11):676-685. doi: 10.1007/s11604-018-0778-4. Epub 2018 Sep 19. PMID 30232584